CLINICAL TRIAL: NCT01231880
Title: School-based Malaria Control: Impact of Intermittent Preventive Treatment on Malaria Morbidity and Cognitive Function in Ugandan School Children
Brief Title: School Based Malaria Control in Ugandan Schoolchildren
Acronym: SBMC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Faculty of Medicine, Dr, Makerere University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MCDC-SBMC
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Malaria
Keywords: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Four monthly IPT (Experimental): IPT give once a school term (every four months)
  Interventions: Drug: Four monthly IPT with dihydroartemisinin Piperaquine (DP)
- Monthly IPT (Experimental): IPT given every month
  Interventions: Drug: Monthly IPT using DP
- Placebo (Placebo Comparator): No active drug in the placebo
  Interventions: Drug: Placebo given every month

INTERVENTIONS:
Drug: Four monthly IPT with dihydroartemisinin Piperaquine (DP) — Given every 4 months (once a school term)
  Other Names: Duocortexin
  Arms: Four monthly IPT
Drug: Monthly IPT using DP — Given every month
  Other Names: Duocortexin
  Arms: Monthly IPT
Drug: Placebo given every month — No active ingredient
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The investigators hypothesize that schoolchildren treated with IPT using DP over one year of follow-up will have a different risk of clinical malaria compared to those treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 6 - 14 years
* Pupils enrolled at participating school
* Willingness of the parent/guardian to provide consent
* Provision of assent by pupil (those above 8 years)

Exclusion Criteria:

* Known allergy or history of adverse reaction to study medications
* Intention of changing of schools during the follow-up period
* History (obtained from the parent/guardian) of any known serious chronic disease requiring frequent medical care

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 740 (Actual)
Dates: Start 2011-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Risk of Clinical Malaria | 1 year
  Fever(temperature greater or equal to 37.5 degrees centigrade or history of fever in past 24 hours) in presence of parasitemia.
Cognitive function tests | 1 year
  Mean score in the cognitive function tests (Raven's Matrices test and Code transmission test)

SECONDARY OUTCOMES:
Risk of parasitemia | 1 year
  presence of asexual parasites on blood smear
Risk of hospital admissions | 1 year
  Admission of any cause
Risk of adverse events | 1 year
  Any untoward medical occurrence in a participant taking study medication
School performance | 1 year
  Average position in class as reported in the end of the year school report
Prevalence of anemia | 1 year
  Proportion of hemoglobin measurements < 10 g/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Joaniter I Nankabirwa, MSc CEB, Principal Investigator — Makerere University Kampala
Locations (1):
- Mulanda Sub-district, Tororo, Uganda, Uganda

REFERENCES:
- [Derived] Nankabirwa JI, Conrad MD, Legac J, Tukwasibwe S, Tumwebaze P, Wandera B, Brooker SJ, Staedke SG, Kamya MR, Nsobya SL, Dorsey G, Rosenthal PJ. Intermittent Preventive Treatment with Dihydroartemisinin-Piperaquine in Ugandan Schoolchildren Selects for Plasmodium falciparum Transporter Polymorphisms That Modify Drug Sensitivity. Antimicrob Agents Chemother. 2016 Sep 23;60(10):5649-54. doi: 10.1128/AAC.00920-16. Print 2016 Oct. PMID 27401569
- [Derived] Nankabirwa JI, Wandera B, Amuge P, Kiwanuka N, Dorsey G, Rosenthal PJ, Brooker SJ, Staedke SG, Kamya MR. Impact of intermittent preventive treatment with dihydroartemisinin-piperaquine on malaria in Ugandan schoolchildren: a randomized, placebo-controlled trial. Clin Infect Dis. 2014 May;58(10):1404-12. doi: 10.1093/cid/ciu150. Epub 2014 Mar 12. PMID 24621953